CLINICAL TRIAL: NCT05116189
Title: A Phase 3, Randomized, Double-Blind Study of Pembrolizumab Versus Placebo in Combination With Paclitaxel With or Without Bevacizumab for the Treatment of Platinum-resistant Recurrent Ovarian Cancer (KEYNOTE-B96/ENGOT-ov65)
Brief Title: Pembrolizumab/Placebo Plus Paclitaxel With or Without Bevacizumab for Platinum-resistant Recurrent Ovarian Cancer (MK-3475-B96/KEYNOTE-B96/ENGOT-ov65)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-B96; MK-3475-B96 (Other: MSD); KEYNOTE-B96 (Other: MSD); ENGOT-ov65 (Other: European Network of Gynaecological Oncological Trial groups); jRCT2051210184 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-506177-35-00 (Registry Identifier: EU CT); U1111-1287-5318 (Registry Identifier: UTN); 2020-005027-37 (EudraCT Number)
Record Dates: First submitted 2021-10-28; First posted 2021-11-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Bevacizumab; Saline Solution; Glucose; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + paclitaxel ± bevacizumab (Experimental): Participants receive pembrolizumab 400 mg via intravenous (IV) infusion for eighteen 6-week cycles (approximately 2 years) PLUS paclitaxel 80 mg/m^2 via IV infusion on Days 1, 8, and 15 of each 3-week cycle until intolerance or disease progression. Participants who experience severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive docetaxel (75 mg/m^2 every 3 weeks [Q3W]) after Sponsor consultation. Participants may also receive bevacizumab 10 mg/kg via IV infusion of each 2-week cycle until intolerance, disease progression, or at the Investigator's discretion.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Bevacizumab; Drug: Docetaxel
- Placebo + paclitaxel ± bevacizumab (Placebo Comparator): Participants receive placebo via IV infusion for eighteen 6-week cycles (approximately 2 years) PLUS paclitaxel 80 mg/m^2 via IV infusion on Days 1, 8, and 15 of each 3-week cycle until intolerance or disease progression. Participants who experience severe hypersensitivity reaction to paclitaxel or an AE requiring discontinuation of paclitaxel may receive docetaxel (75 mg/m^2 every 3 weeks [Q3W]) after Sponsor consultation. Participants may also receive bevacizumab 10 mg/kg via IV infusion of each 2-week cycle until intolerance, disease progression, or at the Investigator's discretion.
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Other: Placebo for pembrolizumab; Drug: Docetaxel

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475,; KEYTRUDA®
  Arms: Pembrolizumab + paclitaxel ± bevacizumab
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: Bevacizumab — IV infusion
  Other Names: AVASTIN®, Zirabev
Other: Placebo for pembrolizumab — IV infusion
  Other Names: normal saline or dextrose
  Arms: Placebo + paclitaxel ± bevacizumab
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®

SUMMARY:
The primary objective is to compare pembrolizumab plus paclitaxel with or without bevacizumab to placebo plus paclitaxel with or without bevacizumab, with respect to progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator. The hypotheses are that pembrolizumab plus paclitaxel with or without bevacizumab is superior to placebo plus paclitaxel with or without bevacizumab, with respect to PFS per RECIST 1.1 as assessed by the investigator for participants with programmed cell death ligand 1 (PD-L1) positive tumors (Combined Positive Score [CPS] ≥1) and that pembrolizumab plus paclitaxel with or without bevacizumab is superior to placebo plus paclitaxel with or without bevacizumab, with respect to PFS per RECIST 1.1 as assessed by the investigator for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Has received 1 or 2 prior lines of systemic therapy for ovarian cancer (OC), including at least 1 prior platinum-based therapy. Participants may have received a prior poly (ADP-ribose) polymerase inhibitor (PARPi), anti-PD-1/anti-PD-L1 therapy, bevacizumab, or hormonal therapy; these will not be considered a separate line of therapy. Any chemotherapy regimen change due to toxicity in the absence of disease progression will be considered part of the same line of therapy.
* Has provided documented informed consent for the study.
* Has radiographic evidence of disease progression within 6 months (180 days) after the last dose of platinum-based chemotherapy for OC (i.e., platinum-resistant disease).
* Is a candidate for paclitaxel chemotherapy (and bevacizumab, if using).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 3 days before randomization.
* For a female participant, she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and uses a contraceptive method that is highly effective (with a failure rate of <1% per year).
* Has radiographically evaluable disease, either measurable or nonmeasurable per RECIST 1.1, as assessed by the local site investigator.
* Archival tumor tissue sample or newly obtained core or incisional/excisional biopsy of a tumor lesion not previously irradiated has been provided.
* Have adequate organ function.

Exclusion Criteria:

* Has nonepithelial cancers, borderline tumors, mucinous, seromucinous that is predominantly mucinous, malignant Brenner's tumor and undifferentiated carcinoma.
* Has primary platinum-refractory disease, defined as disease that has progressed per radiographic imaging while receiving or within 28 days of the last dose of first-line platinum-based therapy.
* Has prior disease progression on weekly paclitaxel alone.
* Has received >2 prior lines of systemic therapy for OC.
* Has received prior systemic anticancer therapy including investigational agents or maintenance therapy (including bevacizumab maintenance therapy), within 4 weeks before randomization.
* Has received prior radiation therapy within 2 weeks of start of study intervention.
* Has not recovered adequately from surgery and/or any complications from the surgery.
* Has received colony-stimulating factors (e.g., granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor,[GM-CSF] or recombinant erythropoietin) within 4 weeks before randomization.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Has received investigational agent or has used an investigational device within 4 weeks prior to study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, paclitaxel, or bevacizumab (if using) and/or any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Participant, in the judgement of the investigator, is unlikely to comply with the study procedures, restrictions, and requirements of the study.
* Has had an allogenic tissue/solid organ transplant.

For bevacizumab treatment

* Has uncontrolled hypertension.
* Has current, clinically relevant bowel obstruction including related to underlying epithelial OC, abdominal fistula or gastrointestinal perforation, intra-abdominal abscess, or evidence of rectosigmoid involvement by pelvic exam.
* Has a history of thrombotic disorders, hemorrhage, hemoptysis, or active gastrointestinal bleeding within 6 months before randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 643 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2028-10-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Investigator | Up to ~38 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on Investigator assessment or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by the Investigator will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~64 months
  OS is defined as the time from the date of randomization to death due to any cause. The OS will be reported for all participants.
PFS per RECIST 1.1 by Blinded Independent Central Review (BICR) | Up to ~38 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review assessment or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by blinded independent central review will be presented.
Number of Participants who Experience an Adverse Event (AE) | Up to ~64 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants who Discontinue Study Treatment due to an AE | Up to ~64 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.
Change From Baseline in Global Health Status/Quality of Life (GHS/Qol) Score (Items 29 and 30) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline and up to ~64 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Time to Deterioration (TTD) in the GHS/Qol Score (Items 29 and 30) Using the EORTC QLQ-C30 | Up to ~64 months
  TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline in GHS (EORTC QLQ-C30 Items 29 and 30) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in GHS score, will be presented. A longer TTD indicates a better outcome.
Change From Baseline in the Abdominal and Gastrointestinal (GI) Symptoms Score (Items 31 to 36) Using the EORTC Quality of Life Questionnaire-Ovarian Cancer (QLQ-OV28) Abdominal/GI Symptom Scale | Baseline and up to ~64 months
  The EORTC QLQ-OV28 is an abdominal and gastrointestinal questionnaire (items 31-36). Participant responses to the question "Did you have abdominal pain ?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in abdominal and gastrointestinal symptoms (EORTC QLQ-LC28 Items 31-36) score will be presented. A lower score indicates a better outcome.
TTD in the Abdominal and GI Symptoms Score (Items 31 to 36) Using the EORTC QLQ-OV28 Abdominal/GI Symptom Scale | Up to ~64 months
  TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline in GHS (EORTC QLQ-C28 Items 31-36) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in GHS score, will be presented. A longer TTD indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (187):
- United States (31):
  - HonorHealth ( Site 0041), Phoenix, Arizona
  - Marin Cancer Care ( Site 0055), Greenbrae, California
  - Pacific Cancer Care ( Site 0028), Monterey, California
  - Eisenhower Medical Center ( Site 0067), Rancho Mirage, California
  - Yale-New Haven Hospital-Smilow Cancer Hospital at Yale-New Haven ( Site 0004), New Haven, Connecticut
  - University of Florida College of Medicine-UF Health Cancer Center/Clinical Trials Office ( Site 0054, Gainesville, Florida
  - Sarasota Memorial Hospital ( Site 0018), Sarasota, Florida
  - Moffitt Cancer Center ( Site 0033), Tampa, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0005), Marietta, Georgia
  - Advocate Medical Group-Oncology ( Site 0049), Park Ridge, Illinois
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0027), Fort Wayne, Indiana
  - St. Vincent Hospital and Health Care Center, Inc ( Site 0032), Indianapolis, Indiana
  - Saint Elizabeth Medical Center Edgewood-Cancer Care Center ( Site 0040), Edgewood, Kentucky
  - WK Physicians Network / Hematology Oncology Associates ( Site 0034), Shreveport, Louisiana
  - Mercy Medical Center - Baltimore-Medical Oncology and Hematology ( Site 0015), Baltimore, Maryland
  - University of Massachusetts Chan Medical School-Division of Gynecologic Oncology ( Site 0003), Worcester, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0007), Hackensack, New Jersey
  - Roswell Park Cancer Institute ( Site 0039), Buffalo, New York
  - Columbia University Medical Center ( Site 0010), New York, New York
  - Novant Health Presbyterian Medical Center ( Site 0029), Charlotte, North Carolina
  - Duke Cancer Institute ( Site 0038), Durham, North Carolina
  - Novant Health Forsyth Medical Center ( Site 0057), Winston-Salem, North Carolina
  - Aultman Hospital-Oncology Clinical Trials ( Site 0009), Canton, Ohio
  - MetroHealth Medical Center-Cancer Care Center ( Site 0047), Cleveland, Ohio
  - Providence Portland Medical Center ( Site 0048), Portland, Oregon
  - University of Pittsburgh Medical Center Magee-Womens Hospital ( Site 0024), Pittsburgh, Pennsylvania
  - Sanford Cancer Center ( Site 0064), Sioux Falls, South Dakota
  - The West Clinic, PLLC dba West Cancer Center ( Site 0058), Germantown, Tennessee
  - Texas Oncology - Dallas (Presbyterian) ( Site 0065), Dallas, Texas
  - Texas Oncology - The Woodlands_Lee ( Site 0043), The Woodlands, Texas
  - Inova Schar Cancer Institute ( Site 0019), Fairfax, Virginia
- Australia (4):
  - Westmead Hospital-Department of Gynaecological Oncology ( Site 0201), Westmead, New South Wales
  - Gallipoli Medical Research Foundation-GMRF CTU ( Site 0202), Brisbane, Queensland
  - Epworth Freemasons ( Site 0204), Melbourne, Victoria
  - St. John of God Subiaco Hospital ( Site 0203), Subiaco, Western Australia
- Belgium (4):
  - Institut Jules Bordet-Medicine Oncology ( Site 0302), Brussels, Bruxelles-Capitale, Region de
  - UZ Gent-Medical oncology ( Site 0301), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0303), Leuven, Vlaams-Brabant
  - AZ Groeninge Campus Kennedylaan-Oncology ( Site 0305), Kortrijk, West-Vlaanderen
- Brazil (6):
  - Hospital Araújo Jorge ( Site 0401), Goiânia, Goiás
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0404), Natal, Rio Grande do Norte
  - ANIMI - Unidade de Tratamento Oncologico ( Site 0408), Lages, Santa Catarina
  - BP - A Beneficencia Portuguesa de São Paulo ( Site 0403), São Paulo, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0405), São Paulo, São Paulo
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA-Pesquisa Clinica HC II ( Site 0402), Rio de Janeiro
- Canada (10):
  - Tom Baker Cancer Center ( Site 0511), Calgary, Alberta
  - BC Cancer Abbotsford ( Site 0512), Abbotsford, British Columbia
  - BC Cancer Victoria ( Site 0513), Victoria, British Columbia
  - Kingston Health Sciences Centre-Kingston General Hospital Si-Oncology and/or Hematology - Gynecolog, Kingston, Ontario
  - Sunnybrook Health Sciences - Odette Cancer Centre ( Site 0508), Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 0501), Montreal, Quebec
  - Jewish General Hospital ( Site 0505), Montreal, Quebec
  - McGill University Health Centre ( Site 0502), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
  - Saskatoon Cancer Center ( Site 0510), Saskatoon, Saskatchewan
- Chile (8):
  - Clínica Puerto Montt ( Site 0601), Port Montt, Los Lagos Region
  - Oncovida ( Site 0603), Santiago, Region M. de Santiago
  - Instituto de Radiomedicina-hemato-oncologia ( Site 0604), Santiago, Region M. de Santiago
  - Clínica Vespucio-Hemato - Ocology ( Site 0607), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Centro del Cáncer ( Site 0609), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0605), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 0602), Temuco, Región de la Araucanía
  - CIDO SpA-Oncology ( Site 0608), Temuco, Región de la Araucanía
- China (29):
  - Anhui Provincial Hospital-Obstetrics and Gynecology ( Site 0709), Hefei, Anhui
  - Beijing Cancer hospital ( Site 0711), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-Gynecological center of tumor ( Site 0702), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0713), Fuzhou, Fujian
  - Lanzhou university second hospital ( Site 0734), Lanzhou, Gansu
  - Zhujiang Hospital ( Site 0739), Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University ( Site 0743), Zhanjiang, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 0717), Nanning, Guangxi
  - Hainan General Hospital ( Site 0736), Haikou, Hainan
  - Henan Cancer Hospital ( Site 0718), Zhengzhou, Henan
  - Wuhan Union Hospital-Medical Oncology ( Site 0735), Wuhan, Hubei
  - Hubei Cancer Hospital-Hubei Cancer Hospital ( Site 0708), Wuhan, Hubei
  - Xiangya Hospital Central South University-Gynecology ( Site 0705), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0704), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Oncology (, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University ( Site 0723), Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital-Oncology Department ( Site 0716), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 0710), Changchun, Jilin
  - Shandong Cancer Hospital-Oncology Department ( Site 0733), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 0731), Linyi, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University ( Site 0715), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center-Gynecologic Oncology Department ( Site 0701), Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital-Gynecology department ( Site 0744), Shanghai, Shanghai Municipality
  - West China Second University Hospital Sichuan University ( Site 0740), Chengdu, Sichuan
  - Tianjin Central Hosptial of Gynecology Obstetrics ( Site 0737), Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital ( Site 0720), Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital-Gynecology Department ( Site 0714), Kunming, Yunnan
  - The Affiliated Women's Hospital of Zhejiang University-Obstetrics and Gynecology ( Site 0741), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Gynecology ( Site 0706), Wenzhou, Zhejiang
- Colombia (5):
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 0808), Medellín, Antioquia
  - Clinica de la Costa LTDA-Clinical Research Oncology & Hematology -Pediatric ( Site 0809), Barranquilla, Atlántico
  - Clínica Universitaria Colombia ( Site 0806), Bogotá, Bogota D.C.
  - Oncologos del Occidente ( Site 0807), Pereira, Risaralda Department
  - Hemato Oncologos SA ( Site 0801), Cali, Valle del Cauca Department
- Aalborg Universitetshospital, Syd ( Site 0901), Aalborg, North Denmark, Denmark
- Turku University Hospital-Department of Obstetrics and Gynecology ( Site 1001), Turku, Southwest Finland, Finland
- France (7):
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital-Institut de cancérologie et hématologi, Brest, Brittany Region
  - Centre François Baclesse-Recherche clinique ( Site 2904), Caen, Calvados
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren-oncologie ( Site 2907), Limoges, Haute-Vienne
  - Institut Curie - site Saint-Cloud ( Site 2909), Saint-Cloud, Hauts-de-Seine
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer-Medical Oncology ( Site 2901), Rennes, Ille-et-Vilaine
  - Centre de Cancérologie du Grand Montpellier ( Site 2908), Montpellier, Languedoc-Roussillon
  - Hôpital privé du Confluent SAS-Service d'oncologie médicale ( Site 2905), Nantes, Loire-Atlantique
- Germany (9):
  - Universitaetsklinikum Erlangen-Klinik für Gynäkologie und Geburtshilfe ( Site 1205), Erlangen, Bavaria
  - Universitätsklinikum Bonn-Gynaecological oncology ( Site 1203), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf-Klinik für Frauenheilkunde & Geburtshilfe ( Site 1204), Düsseldorf, North Rhine-Westphalia
  - Zentrum fuer ambulante gynaekologische Onkologie (ZAGO) ( Site 1207), Krefeld, North Rhine-Westphalia
  - CaritasKlinikum Saarbrücken St. Theresia ( Site 1211), Saarbrücken, Saarland
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Frauenheilkunde und Gebur, Dresden, Saxony
  - Universitätsklinikum Leipzig-Department of Gynecology and Obstetrics ( Site 1213), Leipzig, Saxony
  - Charité Campus Virchow-Klinikum ( Site 1201), Berlin
  - Asklepios Kliniken Hamburg-Asklepios Klinik Barmbek ( Site 1214), Hamburg
- St. James's Hospital-Cancer clinical trials office ( Site 2821), Dublin, Ireland
- Israel (7):
  - Emek Medical Center-Gyn-Onc ( Site 1406), Afula
  - Soroka Medical Center ( Site 1404), Beersheba
  - Rambam Health Care Campus-Gyneco-oncology unit ( Site 1402), Haifa
  - Shaare Zedek Medical Center ( Site 1405), Jerusalem
  - Rabin Medical Center ( Site 1401), Petah Tikva
  - Sheba Medical Center ( Site 1407), Ramat Gan
  - Sourasky Medical Center ( Site 1403), Tel Aviv
- Italy (7):
  - IRCCS - AOU di Bologna-SSD Oncologia medica Addarii ( Site 1501), Bologna, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1503), Milan, Lombardy
  - Ospedale San Gerardo-ASST Monza-Oncologia ( Site 1508), Monza, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 1505), Milan, Milano
  - Ospedale Mauriziano-Ginecologia e Ostetricia ( Site 1507), Turin, Piedmont
  - Azienda Ospedaliera Spedali Civili di Brescia ( Site 1504), Brescia
  - Istituto Europeo di Oncologia IRCCS-Divisione di Ginecologia Oncologica ( Site 1502), Milan
- Japan (13):
  - Aichi Cancer Center Hospital ( Site 1610), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 1609), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 1603), Matsuyama, Ehime
  - Ehime University Hospital ( Site 1606), Tōon, Ehime
  - Kurume University Hospital ( Site 1607), Kurume, Fukuoka
  - Hokkaido University Hospital ( Site 1604), Sapporo, Hokkaido
  - Iwate Medical University Hospital ( Site 1613), Shiwa-gun Yahaba-cho, Iwate
  - Nippon Medical School Musashi Kosugi Hospital ( Site 1614), Kawasaki, Kanagawa
  - Saitama Medical University International Medical Center ( Site 1601), Hidaka-shi, Saitama
  - Shizuoka Cancer Center ( Site 1611), Nakatogari, Shizuoka
  - National Cancer Center Hospital ( Site 1612), Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research ( Site 1605), Koto, Tokyo
  - Osaka International Cancer Institute ( Site 1602), Osaka
- Mexico (5):
  - Investigación Oncofarmacéutica-Investigación clínica ( Site 1706), La Paz, Baja California Sur
  - COI Centro Oncologico Internacional S.A.P.I. de C.V.-Investigation Unit COI ( Site 1703), Mexico City, Mexico City
  - INSTITUTO NACIONAL DE CANCEROLOGIA ( Site 1701), Mexico City, Mexico City
  - iCan Oncology Center Centro Medico AVE ( Site 1704), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 1705), Oaxaca City
- Netherlands (4):
  - Radboudumc ( Site 1802), Nijmegen, Gelderland
  - Leids Universitair Medisch Centrum-Medical Oncology ( Site 1801), Leiden, South Holland
  - Erasmus Medisch Centrum-Medical Oncology ( Site 1803), Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 1804), Utrecht
- Auckland City Hospital ( Site 1901), Auckland, New Zealand
- Universitetssykehuset Nord-Norge HF-Kreftavdelingen ( Site 2001), Tromsø, Troms, Norway
- Poland (8):
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Me-Oddzial Ginekologii Onkologicznej ( Sit, Poznan, Greater Poland Voivodeship
  - Szpital Kliniczny im. Księżnej Anny Mazowieckiej ( Site 2103), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Gynecological Oncology Department ( Sit, Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii-Oddzial Onkologii Ginekologicznej ( Site 2106), Bialystok, Podlaskie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku-Uniwersyteckie Centrum Onkologii ( Site 2104), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Ginekologii, Ginekologii Onkologicznej i Endokrynologii Gi, Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-III Klinika Radioterapii i Chemioterapii ( Site 21, Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 2107), Kielce, Świętokrzyskie Voivodeship
- Russia (5):
  - Chelyabinsk Regional Clinical Oncology Dispensary-Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk, Chelyabinsk Oblast
  - Ogarev Mordovia State University ( Site 2209), Saransk, Mordoviya, Respublika
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF-Chemotherapy #2 ( Site 2211), Moscow, Moscow
  - Moscow City Oncology Hospital #62 ( Site 2214), Krasnogorsk D-t, Moscow Oblast
  - SVERDLOVSK REGIONAL ONCOLOGY DISPENSARY-Oncogynecology Department ( Site 2216), Yekaterinburg, Sverdlovsk Oblast
- South Korea (4):
  - Seoul National University Hospital ( Site 2302), Seoul
  - Severance Hospital, Yonsei University Health System-Gynecologic cancer center ( Site 2303), Seoul
  - Asan Medical Center-Division of Gynecologic Oncology, Dept. of Obstetrics & Gynecology ( Site 2304), Seoul
  - Gangnam Severance Hospital ( Site 2301), Seoul
- Turkey (Türkiye) (8):
  - cukurova universty ( Site 2706), Sarçam, Adana
  - Istanbul Universitesi Cerrahpasa ( Site 2709), Fatih, Istanbul
  - Ege University Medicine of Faculty ( Site 2702), Bornova, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 2704), Adana
  - Ankara University Hospital Cebeci ( Site 2701), Ankara
  - Baskent Universitesi Ankara Hastanesi ( Site 2707), Ankara
  - Bezmialem Vakf Üniversitesi-Oncology ( Site 2705), Istanbul
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma, Istanbul
- United Kingdom (8):
  - Brighton and Sussex University Hospitals NHS Trust ( Site 2803), East Sussex, Brighton And Hove
  - Addenbrooke's Hospital ( Site 2808), Cambridge, Cambridgeshire
  - The Royal Cornwall Hospital ( Site 2804), Truro, Cornwall
  - Westmorland General Hospital ( Site 2815), Kendal, Cumbria
  - Ninewells Hospital and Medical School ( Site 2826), Dundee, Dundee City
  - Leicester Royal Infirmary-HOPE Clinical Trials Unit ( Site 2812), Leicester, England
  - Hammersmith Hospital-Medical Oncology ( Site 2818), London, London, City of
  - Velindre Cancer Centre ( Site 2805), Cardiff

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26220&tenant=MT_MSD_9011